CLINICAL TRIAL: NCT04402463
Title: Effects of Global Postural Exercises Versus Specific Therapeutic Neck Exercises on Pain, Disability, Postural Control, and Neuromuscular Efficiency in Women With Chronic Nonspecific Neck Pain
Brief Title: Effects of Global Postural Exercises Versus Specific Therapeutic Neck Exercises in Chronic Non-specific Neck Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Salamanca (Other)
Collaborators: Instituto Politécnico da Guarda (Other)
Responsible Party: Principal Investigator, Roberto Méndez Sánchez, Professor, University of Salamanca
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 458-2019 USalamanca
Record Dates: First submitted 2020-05-19; First posted 2020-05-26 (Actual); Last update posted 2021-11-02 (Actual); Status verified 2021-10

CONDITIONS: Neck Pain; Chronic Pain
Keywords: Postural Global Reeducation; Exercise; Chronic neck pain; Disability; Postural Control; Cervical muscles
MeSH Terms: conditions — Neck Pain; Chronic Pain; Motor Activity

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: the evaluator (investigator who will carry out the measurements) and the results analysis consultant will be masked.
  After second pre-intervention assessment, the physiotherapist who will apply the interventions will carry out the allocation. Randomization will be done using a computerized randomization system (randomized.com), and concealment of allocation will be ensured by sequentially numbered, opaque, sealed envelopes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GPR Group (Experimental): Global Postural Reeducation with 2 parts in each session:
  1. st: 2 postures in lying position - without gravity load (15 minutes each posture): The aim of these postures is to achieve and maintain postural balance and to stretch the posterior muscle chain. In order to achieve this, specific exercises in the lying position are used. That exercises involve a precise use of contractions, stretch reflexes, light and controlled manual tractions and sustained elongations.
     The maintenance of alignment during posture will be achieved by verbal commands and manual contact of the therapist, guaranteeing the active engagement of patient to reach the correct posture.
  2. st: Standing posture - integration under gravity load (10 minutes): With the participant standing the physiotherapist makes final corrections for postural integration.
  Interventions: Other: Global Postural Reeducation
- Exercise Group (Experimental): Therapeutic exercises. That they will be divided into 3 phases:
  The exercises in these phases will consist in active exercises of the cervical spine and shoulder girdle, motor control exercises, and finally strength and endurance of the cervical flexors and extensors and of the musculature of the shoulder girdle.
  Interventions: Other: Exercise Therapeutic

INTERVENTIONS:
Other: Global Postural Reeducation — The participants will receive treatment along 4 weeks, 2 sessions per week, and 40-45 minutes each session.
  In the treatment 3 of the therapeutic postures of GPR method to will carry out following Souchard's principles of "Global Postural Reeducation"
  Arms: GPR Group
Other: Exercise Therapeutic — The participants will receive treatment along 4 weeks, 2 sessions per week, and 40-45 minutes each session.
  The treatment will be divided into 3 phases, where it initially starts with phase 1 (3 treatments) and progresses to phase 2 (3 treatments) until reaching stage 3 (2 treatments).
  Arms: Exercise Group

SUMMARY:
This study is a randomized, parallel, blinded, clinical trial of treatments. The general objective of this study is to analyze and compare the short-term results, during a 4-week follow-up, of two different treatments in patients with chronic nonspecific neck pain.

The treatments to be applied are Global Postural Reeducation (GPR) and specific therapeutic exercise, applied during 8 treatment sessions in 4 weeks. These treatments will be applied by a physiotherapist with clinical experience in the treatment of cervical pain.

During the study, 4 evaluations will be carried out to assess the effects of the interventions on pain, disability, standing postural control and neuromuscular behavior of the cervical muscles ((1) Baseline (pre-intervention); 2) Second pre-intervention (1 week later); 3) 1st post-intervention after four sessions (1+2 weeks later); 4) Final, 2nd post-intervention (1+4 weeks later))

ELIGIBILITY:
Inclusion Criteria:

* Non-specific chronic neck pain (neck or upper shoulder pain that is not related to a known pathology or injury, with an evolution of at least 12 weeks)

Exclusion Criteria:

* Specific cause of cervical pain (systemic, traumatic, rheumatic pathology, discal pathology,...)
* Central or peripheral neurological signs
* Cognitive impairment to follow instructions during the evaluations or interventions
* History of cervical surgery
* Treatment of physical therapy in the last 3 months
* Pharmacologic treatment during the study

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2021-10-14 (Actual); Study Completion 2021-10-14 (Actual)

PRIMARY OUTCOMES:
Changes in neck pain intensity before, during and after the intervention | 5 weeks. 4 time points: 1) Baseline (pre-intervention); 2) Second pre-intervention (1 week later); 3) 1st post-intervention after four sessions (1+2 weeks later); 4) Final, 2nd post-intervention (1+4 weeks later)
  Numerical Pain Rating Scale (NPRS) will be used. It is a scale used to quantify the patient's pain level on an 11-point numerical scale 0-10 with 0 being "no pain" and 10 being the "worst possible pain."
Changes in disability before, during and after the intervention | 5 weeks. 3 time points: 1) Baseline (pre-intervention); 2) Second pre-intervention (1 week later); 3) Final, 2nd post-intervention (1+4 weeks later)
  The Neck Disability Index (NDI) will be used. It is a modification of the Oswestry Low Back Pain Disability Index. It is a scale used to measure disability associated with cervical pain due to acute or chronic conditions. He has 10 items: 7 related to activities of daily living, 2 related to pain and 1 related to concentration. The test can be interpreted with a maximum score of 50.
  0 - 4 = no disability 5 - 14 = mild 15 - 24 = moderate 25 - 34 = severe above 34 = complete

SECONDARY OUTCOMES:
Changes in Cervical Range of Motion (CROM) before, during and after the intervention | 5 weeks. 4 time points: 1) Baseline (pre-intervention); 2) Second pre-intervention (1 week later); 3) 1st post-intervention after four sessions (1+2 weeks later); 4) Final, 2nd post-intervention (1+4 weeks later)
  The Cervical Range of Motion (CROM) device (Performance Attainment Associates, USA) will be used to measure the cervical range of motion, including flexion, extension, lateral flexion and rotation.
Changes in Pressure Pain Threshold (PPTs) before, during and after the intervention | 5 weeks. 4 time points: 1) Baseline (pre-intervention); 2) Second pre-intervention (1 week later); 3) 1st post-intervention after four sessions (1+2 weeks later); 4) Final, 2nd post-intervention (1+4 weeks later)
  Pressure algometry measurements will be performed with a digital algometer to assess pressure pain thresholds on the trapezius muscles and the spinous process of the 2nd and 6th cervical vertebrae.
Changes in Pain Catastrophizing Scale (PCS) before, during and after the intervention | 5 weeks. 3 time points: 1) Baseline (pre-intervention); 2) Second pre-intervention (1 week later); 3) Final, 2nd post-intervention (1+4 weeks later)
  Pain Catastrophizing Scale (PCS) will be used. People are asked to indicate the degree to which they have the above thoughts and feelings when they are experiencing pain using the 0 (not at all) to 4 (all the time) scale. A total score is yielded (ranging from 0-52).
Changes in Tampa Scale for kinesiophobia (TSK-13) before, during and after the intervention | 5 weeks. 3 time points: 1) Baseline (pre-intervention); 2) Second pre-intervention (1 week later); 3) Final, 2nd post-intervention (1+4 weeks later)
  The Tampa Scale for kinesiophobia (TSK-13) will be used. It is a patient-reported outcome measure designed to help identify kinesiophobia. This version is a 13-item questionnaire aimed at the assessment of fear of movement/re-injury. Each item is provided with a 4-points Likert scale with scoring alternatives ranging from "strongly disagree" [0] to "strongly agree" [4] . This gives a possible total raw score range from 0 to 52.
Changes in Static postural stability before, during and after the | 5 weeks. 3 time points: 1) Baseline (pre-intervention); 2) Second pre-intervention (1 week later); 3) Final, 2nd post-intervention (1+4 weeks later)
  Postural assessment will be examined with the subjects standing on a force platform to evaluate the stabilometry parameters of Center of Pressure (COP) excursions (displacements, velocities, areas and pressures) in different conditions.
Changes in Electromyography parameters of cervical flexor muscles before, during and after the | 5 weeks. 3 time points: 1) Baseline (pre-intervention); 2) Second pre-intervention (1 week later); 3) Final, 2nd post-intervention (1+4 weeks later)
  Surface electromyographic signals will be acquired with electrodes from sternocleidomastoid and anterior scalene muscles.

CONTACTS AND LOCATIONS:
Overall Officials: Roberto Méndez-Sánchez, PhD, Principal Investigator — University of Salamanca
Locations (2):
- Instituto Politécnico da Guarda, Guarda, Portugal
- University of Salamanca, Salamanca, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mendes-Fernandes T, Puente-Gonzalez AS, Marquez-Vera MA, Vila-Cha C, Mendez-Sanchez R. Effects of Global Postural Reeducation versus Specific Therapeutic Neck Exercises on Pain, Disability, Postural Control, and Neuromuscular Efficiency in Women with Chronic Nonspecific Neck Pain: Study Protocol for a Randomized, Parallel, Clinical Trial. Int J Environ Res Public Health. 2021 Oct 12;18(20):10704. doi: 10.3390/ijerph182010704. PMID 34682453